CLINICAL TRIAL: NCT00697658
Title: INVega Is Studied In an Observational Design in the Netherlands
Brief Title: INVISION - An Observational Study to Explore Effectiveness, Tolerability and Safety of Paliperidone ER in Patients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR014788; R076477SCH4017
Record Dates: First submitted 2008-04-11; First posted 2008-06-16 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Schizophrenia
Keywords: Paliperidone ER; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — 6 mg tablet once daily, variable treatment length.

SUMMARY:
The purpose of this study is to explore efficacy, tolerability and safety of paliperidone Extended Release (ER) in 250 schizophrenia patients who started treatment with paliperidone ER in a naturalistic setting.

DETAILED DESCRIPTION:
This is an observational, prospective, multicenter 6-month study to explore efficacy, tolerability and safety of paliperidone Extended Release (ER) in 250 schizophrenia patients who started treatment with paliperidone ER in a naturalistic setting. The primary objective is to explore changes in Clinical Global Impression of Severity (CGI-S) score from baseline up to 26 weeks, in subgroups of schizophrenia patients who started treatment with paliperidone ER. Secondary objectives are: 1) To explore changes in mental health and social functioning based on routine outcome assessments in the Netherlands, the Health of the Nation Outcome Scales (HoNOS) and Global Assessment of Functioning (GAF), in schizophrenia patients who started treatment with paliperidone ER ; 2) To explore changes in patient's satisfaction with treatment, changes in number of ambulant contacts, changes in body weight, changes in concomitant therapy and to explore adverse events in schizophrenia patients who started treatment with paliperidone ER; and to explore possible association between CGI-S, GAF and HoNOS.

The patients will receive paliperidone ER (6 mg, 9 mg or other dosages as directed on the label) once daily for the period of 6 month. Which dosage of paliperidone ER the patients receive will be at the discretion of the investigator and according the Summary of Product Characteristics (SmPC). Because the study is observational, dosage, administration and duration of treatment is at discretion of treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets the DSM-IV criteria for schizophrenia
* Switched to or started on paliperidone ER, not longer than two weeks ago
* In 24 hours before initiation of paliperidone ER treatment, CGI-S, patient satisfaction with treatment, concomitant therapy, body weight, GAF and HoNOS data are available
* Patient or legal representative has signed the informed consent form within two weeks after starting treatment with paliperidone ER

Exclusion Criteria:

* No use of paliperidone ER, clozapine, any conventional depot neuroleptic or long acting atypical antipsychotic drugs during 3 months before starting paliperidone ER
* No participation in an investigational drug trial in 30 days prior to starting paliperidone ER
* No history of neuroleptic malignant syndrome
* No known hypersensitivity to paliperidone ER or risperidone
* No patients hospitalized for a period longer than 12 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Schizophrenia patients meeting DSM-IV criteria receiving paliperidone ER, as part of the common practice of participating physicians. Patients may enter the study as soon as their paliperidone ER treatment starts or when it has been less than 14 days after their treatment start.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2008-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in CGI-S score at the end of the study | Week 26 or drop out visit

SECONDARY OUTCOMES:
Change in Health of the Nation Outcome Scales (HoNOS) | Week 26 or drop out visit
Change in GAF score | Week 26 or drop out visit
Patient satisfaction with treatment | Week 26 or drop out visit

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag B.V. Clinical Trial, Study Director — Janssen-Cilag B.V.
Locations (17):
- Netherlands (17):
  - Alphen aan den Rijn
  - Amersfoort
  - Amsterdam
  - Beverwijk
  - Deventer
  - Echt
  - Enschede
  - Geldrop
  - Heerde
  - Heerenveen
  - Hoorn
  - Kampen
  - Nijmegen
  - Purmerend
  - Roermond
  - Vlaardingen
  - Zwolle